CLINICAL TRIAL: NCT02495181
Title: A Randomized, Double-masked, Sham-controlled Phase 4 Study of the Efficacy, Safety, and Tolerability of IV Aflibercept Monotherapy Compared to Aflibercept With Adjunctive Photodynamic Therapy in Patients With PCV.
Brief Title: Randomized, Double-masked, Sham-controlled Phase 4 Study, Efficacy, Safety, and Tolerability of Intravitreal Aflibercept Monotherapy Compared to Aflibercept With Adjunctive Photodynamic Therapy in Patients With Polypoidal Choroidal Vasculopathy
Acronym: ATLANTIC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Association for Innovation and Biomedical Research on Light and Image (Other)
Collaborators: European Vision Institute Clinical Research Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ECR-AMD-2015-09
Record Dates: First submitted 2015-03-23; First posted 2015-07-13 (Estimated); Last update posted 2020-01-10 (Actual); Status verified 2019-02

CONDITIONS: Polypoidal Choroidal Vasculopathy
MeSH Terms: conditions — Polypoidal Choroidal Vasculopathy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aflibercept Monotherapy (Sham Comparator): IVT Aflibercept 2 mg + Sham PDT
  Interventions: Drug: Intravitreal Aflibercept
- Aflibercept + verteporfin PDT (Active Comparator): IVT Aflibercept 2 mg + Verteporfin PDT
  Interventions: Drug: Intravitreal Aflibercept

INTERVENTIONS:
Drug: Intravitreal Aflibercept
  Other Names: standard photodynamic therapy (PDT)

SUMMARY:
The purpose of this study is to compare the efficacy and safety of intravitreal Aflibercept monotherapy with the efficacy and safety of combined treatment with Aflibercept plus standard photodynamic therapy (PDT) with Verteporfin in age-related macular degeneration (AMD) patients with polypoidal choroidal vasculopathy (PCV).

DETAILED DESCRIPTION:
To compare the efficacy and safety of intravitreal Aflibercept monotherapy with the efficacy and safety of combined treatment with Aflibercept associated with standard photodynamic therapy (PDT) with Verteporfin in age-related macular degeneration (AMD) patients with polypoidal choroidal vasculopathy (PCV) in a proof concept study and to identify genetic biomarkers for the diagnosis and treatment response of PCV in Caucasians.

ELIGIBILITY:
Inclusion Criteria:

* Either gender and Age ≥ 50.
* Naïve PCV patients.
* Confirmed diagnosis of symptomatic macular PCV in the study eye.
* Greatest linear dimension of the lesion of < 5400 mm, assessed by ICG angiography.
* BCVA at study entry of 25 to 80 letters (Snellen Equivalent 20/320 to 20/25).
* Lesion size in the study eye at study entry:
* Presence of PCV assessed by the Central Reading Centre based on ICG with active polyps with or without abnormal vascular network.
* Women must be using effective contraception, be post-menopausal for at least
* months prior to trial entry, or surgically sterile.
* Ability to provide written informed consent.
* Ability to return for all study visits.

Exclusion Criteria:

* Active inflammation or infection in the study eye.
* Uncontrolled intraocular pressure in the study eye.
* Ocular condition in the study eye which may impact vision and confound study outcomes (e.g. vitreomacular traction, epirretinal membrane with BCVA impact, ocular inflammation, retinal vascular diseases like diabetic retinopathy or diabetic macular edema).
* Presence of centromacular scarring or atrophy indicating irreversible BCVA loss.
* Prior treatment of the study eye with anti-VEGF therapy or systemic use of anti-VEGF products within 3 months prior to the study entry.
* Previous vitrectomy, macular laser treatment, PDT, or intraocular steroids in the study eye.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-11-23 (Actual); Primary Completion 2017-08-22 (Actual); Study Completion 2019-12-17 (Actual)

PRIMARY OUTCOMES:
Change in Best Corrected Visual Acuity (BCVA) | from Baseline (Week 0) to Week 52.
  Unit of Measure: [Letters]
Polyps regression | from Baseline (W0) to Week 52.
  Unit of Measure: [Yes, No]

SECONDARY OUTCOMES:
Polyps regression, assessed by Indocyanine Green Angiography (ICGA); | from Baseline (W0) to Week 16
  Unit of Measure: [Yes, No]
Presence of active polyps, assessed by Indocyanine Green Angiography (ICGA); | from Baseline (W0) to Week 52
  Unit of Measure: [Yes, No]
Presence of leakage based on fluorescein angiography (FA) | from Baseline (W0) to Week 52
  Unit of Measure: [Yes, No]
Change in the Subfield Central Retinal Thickness (CRT), assessed by Spectral Domain-Optical Coherence Tomography (SD-OCT); | from Baseline (W0) to Week 52
  Unit of Measure: [µm]
Presence of fluid assessed on Spectral Domain-Optical Coherence Tomography (SD-OCT) at Week 52; | from Baseline (W0) to Week 52
  Unit of Measure: [Yes, No]
Total number of treatments with Aflibercept; | from Baseline (W0) to Week 52
  Unit of Measure: [#]
Frequency and severity of ocular and non-ocular adverse events over time. | from Baseline (W0) to Week 52
  Unit of Measure: [Mild, Moderate, Severe]

CONTACTS AND LOCATIONS:
Overall Officials: Rufino Silva, PhD, Principal Investigator — Association for Innovation and Biomedical Research on Light and Image
Locations (13):
- Portugal (9):
  - Hospital de Braga, Braga
  - AIBILI - Centro de Ensaios Clínicos, Coimbra
  - Espaço Médico de Coimbra, Coimbra
  - Centro Hospitalar de Leiria, Leiria
  - IRL - Instituto de Retina e Diabetes de Lisboa, Lisbon
  - Centro Hospitgalar de Lisboa Norte, EPE - Hospital de Santa Maria, Lisbon
  - Instituto de Oftalmologia Dr. Gama Pinto, Lisbon
  - Centro Hospitalar do Porto- Hospital de Santo António, Porto
  - Centro Hospitalar de São João, EPE - Serviço de Oftalmologia, Porto
- Spain (4):
  - Bellvitge University Hospital, Barcelona
  - Instituto de Microcirugia Ocular, Barcelona
  - Vall d'Hebron Hospital, Barcelona
  - Hospital Insular de Gran Canaria, Las Palmas

REFERENCES:
- [Derived] Silva R, Arias L, Nunes S, Farinha C, Coimbra R, Marques JP, Cachulo ML, Figueira J, Barreto P, Madeira MH, Pires I, Sousa JC, Distefano L, Rosa P, Carneiro A, Vaz-Pereira S, Meireles A, Cabrera F, Bures A, Mendonca L, Fernandez-Vega-Sanz A, Barrao S, Koh A, Cheung CMG, Cunha-Vaz JG, Murta J; EVICR.net ATLANTIC Study Group. Efficacy and Safety of Intravitreal Aflibercept Treat and Extend for Polypoidal Choroidal Vasculopathy in the ATLANTIC Study: A Randomized Clinical Trial. Ophthalmologica. 2022;245(1):80-90. doi: 10.1159/000518235. Epub 2021 Jul 13. PMID 34348351
- [Derived] Marques JP, Farinha C, Costa MA, Ferrao A, Nunes S, Silva R. Protocol for a randomised, double-masked, sham-controlled phase 4 study on the efficacy, safety and tolerability of intravitreal aflibercept monotherapy compared with aflibercept with adjunctive photodynamic therapy in polypoidal choroidal vasculopathy: the ATLANTIC study. BMJ Open. 2017 Aug 28;7(8):e015785. doi: 10.1136/bmjopen-2016-015785. PMID 28851779